CLINICAL TRIAL: NCT00946998
Title: Randomized Trial of Sertraline Treatment of Depression in Chronic Kidney Disease
Brief Title: Chronic Kidney Disease Antidepressant Sertraline Trial
Acronym: CAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Texas Southwestern Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-008-09S; 1I01CX000217-01 (NIH); 1R01DK085512-01A1 (NIH)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Disease; Depression
Keywords: Chronic Kidney Disease; Depression; Antidepressants; randomized controlled trial; treatment; Sertraline
MeSH Terms: conditions — Renal Insufficiency, Chronic; Depression | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sertraline (Active Comparator): Patients with predialysis Chronic Kidney Disease stages 3-5 and with major depressive episode
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Patients with predialysis Chronic Kidney Disease stages 3-5 and with major depressive episode
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Sertraline — Sertraline is a serotonin-selective reuptake inhibitor (SSRI) used to treat major depression. Dosage will begin at 50 mg/d and will be escalated by 50 mg increments every 2 weeks to a maximum of 200 mg/d
  Arms: Sertraline
Drug: placebo — Placebo tablet will be identical and matched to sertraline tablet.
  Arms: Placebo

SUMMARY:
This is a randomized double-blinded placebo-controlled trial to see if treatment with sertraline as compared with placebo tablets will improve depression symptoms in patients with chronic kidney disease who have not yet started dialysis or received a kidney transplant. The investigators will also investigate whether sertraline treatment will improve quality of life and whether it is safe to use in patients with kidney disease. The study subject will be randomly assigned to take either sertraline or a placebo tablet for 12 weeks.

DETAILED DESCRIPTION:
This is a randomized double-blinded placebo-controlled trial of adults with predialysis stages 3-5 Chronic Kidney Disease and Major Depressive Episode. Subjects will be randomized in a double-blind fashion to placebo or sertraline (beginning at 50 mg/d and escalated by 50 mg increments every 2 weeks to a maximum of 200 mg/d) and followed for 12 weeks. The primary outcome is to investigate if treatment with sertraline, as compared with placebo, results in an improvement in depression symptom severity as measured by the Quick Inventory of Depressive Symptomatology Clinician Rated (QIDS-C-16) score. Secondary outcomes include whether sertraline, as compared with placebo, improves overall function and quality of life and whether it will result in more serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged greater than 21 years.
* Predialysis stages 3, 4 or 5 CKD.
* Current Major Depressive Episode.
* QID-C-16 score of 11.
* Able to understand and sign informed consent.

Exclusion Criteria:

* No healthcare power of attorney to sign informed consent.
* Unwilling or unable to participate.
* Kidney transplant recipient.
* Initiated on maintenance dialysis
* Significant hepatic dysfunction or liver enzyme abnormalities 3 times the upper limits of normal.
* Terminal chronic obstructive pulmonary disease or cancer.
* Recent history of active bleeding, such as gastrointestinal bleeding requiring hospitalization 3 months prior
* Current use of class I anti-arrhythmic medications.
* Use of pimozide, MAO inhibitors, reserpine, guanethidine, cimetidine or methyldopa; tri-cyclic anti-depressants, neuroleptics or anti-convulsants, excluding gabapentin
* Use of other serotonergic drugs or supplements such as triptans, tramadol, linezolid, tryptophan, and St. John's Wort.
* Ongoing use of anti-depressants
* Past treatment failure on Sertraline
* Initiation of psychotherapy for depression in the 3 months prior to study entry
* Alcohol or substance abuse or dependence that requires acute detoxification at study entry
* Present or past psychosis or Bipolar I or II disorder
* Dementia or a Mini-Mental State Examination score of <23
* Suicidal ideation
* Pregnancy, lactation and women of childbearing potential not using adequate contraception

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2010-02-08 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Hedayati, MD MHS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jain N, Trivedi MH, Rush AJ, Carmody T, Kurian B, Toto RD, Sarode R, Hedayati SS. Rationale and design of the Chronic Kidney Disease Antidepressant Sertraline Trial (CAST). Contemp Clin Trials. 2013 Jan;34(1):136-44. doi: 10.1016/j.cct.2012.10.004. Epub 2012 Oct 22. PMID 23085503
- [Result] Hedayati SS, Gregg LP, Carmody T, Jain N, Toups M, Rush AJ, Toto RD, Trivedi MH. Effect of Sertraline on Depressive Symptoms in Patients With Chronic Kidney Disease Without Dialysis Dependence: The CAST Randomized Clinical Trial. JAMA. 2017 Nov 21;318(19):1876-1890. doi: 10.1001/jama.2017.17131. PMID 29101402
- [Derived] Gregg LP, Carmody T, Le D, Bharadwaj N, Trivedi MH, Hedayati SS. Depression and the Effect of Sertraline on Inflammatory Biomarkers in Patients with Nondialysis CKD. Kidney360. 2020 Apr 13;1(6):436-446. doi: 10.34067/KID.0000062020. eCollection 2020 Jun 25. PMID 35368605
- [Derived] Jain N, Wan F, Kothari M, Adelodun A, Ware J, Sarode R, Hedayati SS. Association of platelet function with depression and its treatment with sertraline in patients with chronic kidney disease: analysis of a randomized trial. BMC Nephrol. 2019 Oct 29;20(1):395. doi: 10.1186/s12882-019-1576-7. PMID 31664940

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 102 | 99
Received Treatment as Randomized | 102 | 99
Completed | 97 | 96
Not Completed | 5 | 3
Not completed — Exited prior to first outcome assessment | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 97 | 96 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (14.5) | 59.1 (12.2) | 58.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 52
  Male | 74 | 67 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 14 | 35
  Not Hispanic or Latino | 76 | 82 | 158
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 55 | 111
  White | 41 | 40 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 97 | 96 | 193
Chronic Kidney Disease Stage [Count of Participants; unit: Participants] — Chronic kidney disease stages were categorized as follows: stage 3, estimated glomerular filtration rate (eGFR) of 30 to 59 mL/min/1.73 m^2; stage 4, eGFR of 15-29; and stage 5, eGFR<15, but not dialysis-dependent.
  Participants
    CKD Stage 3 | 46 | 44 | 90
    CKD Stage 4 | 34 | 36 | 70
    CKD Stage 5 | 17 | 16 | 33
Diabetes Mellitus [Count of Participants; unit: Participants] | 58 | 55 | 113
Estimated glomerular filtration rate [Median (Inter-Quartile Range); unit: mL/min/1.73 m^2] | 27.0 [18.0 to 35.0] | 27.5 [17.0 to 38.5] | 27.5 [17.0 to 37.0]
16-item Quick Inventory of Depression Symptomatology Clinician-rated Score [Mean (Standard Deviation); unit: units on a scale] — The 16-item Quick Inventory of Depression Symptomatology measures depressive symptom severity. The range of final score is 0-27, with higher scores indicating more severe depression. A score of 0-5 corresponds to normal affect, 6-10 to mild, 11-15 to moderate, 16-20 to severe, and 21 to very severe depression.
  units on a scale | 14.0 (2.4) | 14.1 (2.4) | 14.0 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Exit in Depression Symptom Severity as Measured by the QIDS-C-16 Score.
Description: The score range is 0 to 27; higher scores indicate more severe depression; a score of 0 to 5 corresponds to a normal affect; 6 to 10 to a mild affect; 11 to 15 to a moderate affect; 16 to 20 to a severe affect; and 21 or greater to very severe depression.
Time Frame: baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 97 | 96
units on a scale | -4.1 [-5.1 to -3.1] | -4.2 [-5.0 to -3.5]
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority; p = 0.82, Mixed Models Analysis

2. Secondary Outcome: Response to Treatment Defined as a Decline of 50% in the Baseline QIDS-C-16 Score and Remission of Depression Defined as a QIDS-C-16 Score of 5
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Measure: Number; unit: participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 97 | 96
participants
  Response (>/=50% decline in score) | 31 | 24
  Remission (score =/<5) | 15 | 14
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority; p = 0.28, Mixed Models Analysis — Represents the response outcome
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Test type: Superiority; p = 0.86, Mixed Models Analysis — Represents remission outcome

3. Secondary Outcome: Change From Baseline to Exit in Overall Function as Assessed by the Work and Social Adjustment Scale
Description: Each item is rated on a 0 to 8 Likert scale with 0 indicating no impairment and 8 indicating severe impairment and a total score range of 0 to 40.
Time Frame: baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 97 | 96
units on a scale | -5.0 [-7.6 to -2.5] | -3.2 [-5.8 to -0.7]
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority; p = 0.32, Mixed Models Analysis

4. Secondary Outcome: Change in Quality of Life From Baseline to Exit in the Kidney Disease Quality of Life -Short Form, Version 1.3, Patient-reported Overall Health.
Description: Raw scores from version 1.3 were transformed to a scale from 0 to 100, in which higher numbers signify more favorable quality of life.
Time Frame: baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 97 | 96
units on a scale | 0.0 [-10.0 to 10.0] | 0.0 [0.0 to 10.0]
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority; p = 0.61, Mixed Models Analysis

5. Secondary Outcome: Serious Adverse Events During the 12 Week Study Duration.
Description: death, dialysis initiation, hospitalizations, or bleeding requiring transfusion
Time Frame: during 12 week study duration
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 97 | 96
Participants
  Death | 0 | 0
  Dialysis initiation | 7 | 5
  Hospitalization other than dialysis initiation | 8 | 7
  acute suicidal intent | 0 | 1
  bleed with transfusion or hospitalization | 2 | 2
Statistical Analysis 1: Comparison: Sertraline vs Placebo; Test type: Superiority; p > .99, Chi-squared — For death
Statistical Analysis 2: Comparison: Sertraline vs Placebo; Test type: Superiority; p = 0.77, Chi-squared — For comparison of dialysis initiation between groups
Statistical Analysis 3: Comparison: Sertraline vs Placebo; Test type: Superiority; p > 0.99, Chi-squared — Hospitalization other than dialysis initiation
Statistical Analysis 4: Comparison: Sertraline vs Placebo; Test type: Superiority; p = 0.5, Chi-squared — For comparison of acute suicidal intent
Statistical Analysis 5: Comparison: Sertraline vs Placebo; Test type: Superiority; p > 0.99, Chi-squared — For comparison of bleeding requiring blood transfusion or hospitalization

ADVERSE EVENTS:
Time Frame: 12 weeks of randomized study duration.
Arm/Group | Sertraline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/96
Serious Adverse Events (participants affected / at risk) | 13/97 | 13/96
Other Adverse Events (participants affected / at risk) | 55/97 | 35/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (N=97) | Placebo (N=96)
Dialysis initiation (Renal and urinary disorders) | 7 | 5 — Initiation of chronic dialysis
Hospitalization other than for dialysis initiation (General disorders) | 8 | 7
acute suicidal intent (Psychiatric disorders) | 0 | 1
Bleeding requiring a blood transfusion or hospitalization (Blood and lymphatic system disorders) | 2 | 2
stroke (Nervous system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (N=97) | Placebo (N=96)
Nausea, indigestion, or vomiting (Gastrointestinal disorders) | 22 | 10
Diarrhea (Gastrointestinal disorders) | 13 | 3
anorexia (Gastrointestinal disorders) | 1 | 1
Increased appetite (Gastrointestinal disorders) | 1 | 2
Insomnia (General disorders) | 7 | 10
Somnolence (General disorders) | 9 | 5
Decreased memory or confusion (Nervous system disorders) | 2 | 3
Dizziness, syncope, or fall (General disorders) | 8 | 4
Anxiety, irritability, or agitation (Psychiatric disorders) | 7 | 4
Tremor (Nervous system disorders) | 3 | 1
Headache (General disorders) | 6 | 4
Dry mouth (General disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Decrease libido or erectile dysfunction (Reproductive system and breast disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No